CLINICAL TRIAL: NCT02522078
Title: Dry vs Wet Misoprostol for Cervical Dilation in First Trimester Abortion - A Clinical Trial
Brief Title: Dry vs Wet Misoprostol for Cervical Dilation in First Trimester Abortion
Acronym: MisoWet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0115
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Abortion Early
Keywords: misoprostol; abortion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Misoprostol (Active Comparator): 400 µg of dry misoprostol
  Interventions: Drug: dry misoprostol
- Wet misoprostol (Experimental): 400 µg of wet misoprostol
  Interventions: Drug: wet misoprostol

INTERVENTIONS:
Drug: dry misoprostol — 400 µg of dry misoprostol will be introduced into the vaginal fornices 3 or more hours before uterine evacuation
  Arms: Dry Misoprostol
Drug: wet misoprostol — 400 µg of wet misoprostol will be introduced into the vaginal fornices 3 or more hours before uterine evacuation
  Arms: Wet misoprostol

SUMMARY:
This study aims to verify whether the moisture of 400 µg of misoprostol pre uterine evacuation increases the dilatation of uterine cervix compared to dry misoprostol

DETAILED DESCRIPTION:
Misoprostol is the most widely used drug for abortion due to its low cost, stability and easy to use regimen. Nevertheless, there is a debate whether the administration of dry misoprostol has similar effects compared to wet pill. It would be necessary to undertake a clinical trial to evaluate which regimen (dry or wet) offers a better cervical dilation pre uterine evacuation. The primary objective of this study is to compare the degree of cervical dilatation pre-uterine evacuation in subject that received 400 µg of dry or wet misoprostol 3 or more hours before the procedure. Secondary objective is to verify whether there is a correlation between vaginal pH (<5 / ≥5) and the degree of cervical dilation (≥8mm / <8mm) with the use of wet or dry misoprostol. Women will be randomized to one of the two groups: dry or wet misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Women with abortion (less than 12 weeks of pregnancy)

Exclusion Criteria:

* congestive heart failure
* chronic pulmonary disease
* hypovolemic shock
* twins
* Marfan syndrome
* septic abortion (fever, pus , leukocytosis >14,000)
* known allergies to misoprostol
* blood dyscrasia
* open cervical (≥ 1cm)
* use of intrauterine device

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cervical dilation | 3 to 4 hours after putting misoprostol into the vagina
  Cervical dilation will be measure with Karman cannulas

SECONDARY OUTCOMES:
Vaginal acidity - hydrogen ion concentration | within 2 min before putting the misoprostol into the vagina
  at the moment of the introduction of misoprostol into the vagina

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WHO. The Prevention and management of unsafe abortion: report of a technical working group, Geneva, 12-15 April 1992. 1993
- [Background] Regan L, Rai R. Epidemiology and the medical causes of miscarriage. Baillieres Best Pract Res Clin Obstet Gynaecol. 2000 Oct;14(5):839-54. doi: 10.1053/beog.2000.0123. PMID 11023804
- [Background] Grimes DA, Benson J, Singh S, Romero M, Ganatra B, Okonofua FE, Shah IH. Unsafe abortion: the preventable pandemic. Lancet. 2006 Nov 25;368(9550):1908-19. doi: 10.1016/S0140-6736(06)69481-6. PMID 17126724
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Neilson JP, Gyte GM, Hickey M, Vazquez JC, Dou L. Medical treatments for incomplete miscarriage. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD007223. doi: 10.1002/14651858.CD007223.pub3. PMID 23543549
- [Background] Fong YF, Singh K, Prasad RN. A comparative study using two dose regimens (200 microg or 400 microg) of vaginal misoprostol for pre-operative cervical dilatation in first trimester nulliparae. Br J Obstet Gynaecol. 1998 Apr;105(4):413-7. doi: 10.1111/j.1471-0528.1998.tb10126.x. PMID 9609268